CLINICAL TRIAL: NCT03498183
Title: Value of the Combination Ultrasonography With Ti-RADS Score / Dual Tracer Scintigraphy MIBI-Tc99m/Iodine-123 in the Detection of Malignancy of Thyroid Nodules (Sup or Egal to 15 mm) Classified Bethesda III or IV on Cytology
Brief Title: Value of the Combination Ultrasonography With Ti-RADS Score / Dual Tracer Scintigraphy MIBI-Tc99m/Iodine-123 in the Detection of Malignancy of Thyroid Nodules (≥15 mm) Classified Bethesda III or IV on Cytology
Acronym: MIBI-THYR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC18_0052
Record Dates: First submitted 2018-03-29; First posted 2018-04-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Malignancy of Thyroid Nodules
MeSH Terms: interventions — Iodine-123

STUDY DESIGN:
Intervention Model Description: All the patients will have the scintigraphie with MIBI-Tc99m/Iodine-123
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARM experimental (Experimental): All the patients will have MIBI-Tc99m/Iodine-123 . Following the injections they will have a scintigraphy.
  Interventions: Drug: MIBI-Tc99m/Iodine-123

INTERVENTIONS:
Drug: MIBI-Tc99m/Iodine-123 — Following the injection of MIBI-Tc99m/Iodine-123 , the patients will have a scintigraphy.

SUMMARY:
The main objective of the study is to show that the addition of ultrasonography to the dual tracer scintigraphy MIBI-Tc99m/Iodine-123 will increase (at least +5%) the negative predictive value compared to the dual tracer scintigraphy alone in detection of malignancy in thyroid nodules ≥15 mm classified as Bethesda III-IV on cytology.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years with a thyroid nodule ≥15 mm (maximal diameter measured on US) with a Bethesda class III or IV (FNA less than 6 months before the surgery).
* Given signed, written informed consent
* Affiliation to a social security system.
* Neither-pregnant nor breast-feeding women.
* Use of efficient contraception for patient with pregnancy potential (if needed).

Exclusion Criteria:

* Underage and adults under guardianship.
* Pregnant, without efficient contraception (if needed) or breast feeding women.
* Administration of iodinated contrast in the previous 3 weeks.
* Contraindication to scintigraphy or to Iodine123/ MIBI 99Tc administration
* Treatment containing iodine (i.e. : Amiodarone)
* Hypo or hyperthyroidism treated or not.
* Nodules inferior 15 mm.
* Refusal to sign the consent.
* Refusal of surgical treatment or contraindication for surgery or anesthesia
* Morbid obesity (BMI Superior 40 kg/m2).
* Hyperparathyroidism.
* History of cervicotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Addition of ultrasonography to the dual tracer scintigraphy MIBI-Tc99m/Iodine-123 will increase the negative predictive value compared to the dual tracer scintigraphy alone. | Month 36
  Scintigraphy MIBI-Tc99m/Iodine-123

SECONDARY OUTCOMES:
Evaluation of the correlation between dual scintigraphy (MIBI/Iodine-123) and cervical ultrasonography (with Ti-RADS score). | Month 36
  Spearman's correlation coefficient between measures obtained using dual scintigraphy (MIBI/Iodine-123) and cervical ultrasonography (with Ti-RADS score).
Evaluation of diagnostics properties of MIBI/Iodine-123 scintigraphy for detection of thyroid malignancy. | Month 36
  Estimation of the sensitivity of MIBI/Iodine-123 scintigraphy for detection of thyroid malignancy.
Evaluation of diagnostics properties of MIBI/Iodine-123 scintigraphy for detection of thyroid malignancy. | Month 36
  Estimation of the specificity value of MIBI/Iodine-123 scintigraphy for detection of thyroid malignancy.
Evaluation of diagnostics properties of MIBI/Iodine-123 scintigraphy for detection of thyroid malignancy. | Month 36
  Estimation of the positive predictive value of MIBI/Iodine-123 scintigraphy for detection of thyroid malignancy.
Evaluation of diagnostics properties of Ti-RADS scoring. | Month 36
  Quality of life measured using the scores of the SF36 questionnaire
Evaluation of diagnostics properties of Ti-RADS scoring. | Month 36
  Quality of life measured using an evaluation of the voice measured using a specific autoquestionnaire
Evaluation of diagnostics properties of Ti-RADS scoring. | Month 36
  Quality of life measured using the scores of EQ-5D questionnaire
Evaluation of diagnostics properties of the best combination of the scintigraphic values (intensity of MIBI and Iodine uptakes) to improve the diagnostic properties. | Month 36
  Research of the best thresholds on scintigraphic values (intensity of MIBI and Iodine uptakes) to improve the diagnostic properties (details of scores are given in "5.3.3. Role of Nuclear Medicine Physician")
Evaluation of the MIBI washout | Month 36
  MIBI washout estimated using the percentage reduction value of mean MIBI uptake between early (10 min) and late (>60 min) scans
Cost-effectiveness analysis (economic efficiency) at 10 years comparing the systematic surgery strategy to the non-systematic strategy guided by imagery. | Month 36
  Incremental cost-effectiveness ratio (cost per Quality-Adjusted Life-Year, QALY) of the comparison between the systematic surgery strategy to the non-systematic surgery strategy guided by imagery over a 10 years' time horizon.
Cost-effectiveness analysis (economic efficiency) at 10 years comparing the systematic surgery strategy to the non-systematic strategy guided by imagery. | year 10
  Incremental cost-effectiveness ratio (cost per Quality-Adjusted Life-Year, QALY) of the comparison between the systematic surgery strategy to the non-systematic surgery strategy guided by imagery over a 10 years' time horizon.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - hopital Avicenne, Bobigny
  - CHU, Lille
  - CHU, Limoges
  - Hospices Civils, Lyon
  - CHU, Nantes
  - Assistance publique des Hôpitaux de Paris, Paris
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: Undecided